CLINICAL TRIAL: NCT07397676
Title: Effects of Breathing Technique Training and Physical Activity Counseling on Quality of Life, Symptoms, Asthma Control, and Physical Activity in Children and Adolescents With Asthma: A Randomized Controlled Trial
Brief Title: Quality of Life - Effects of a Physical Therapy Intervention to for Children and Adolescents With Asthma
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Helene Alexanderson, Associate professor, PhD, RPT, Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KarolinskaUH; F2020-0009 (Other Grant/Funding Number: Swedish Asthma and Allergy Society); 2023-01011 (Other Grant/Funding Number: Promobilia Foundation)
Record Dates: First submitted 2026-02-02; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Paediatric Asthma; Paediatric Dysfunctional Breathing
Keywords: Physical activity; Breathing retraining; Quality of life; Dysfunctional breathing
MeSH Terms: conditions — Motor Activity | interventions — Breathing Exercises

STUDY DESIGN:
Intervention Model Description: Four weeks of randomiazed controlled interventions vs control intervention with an additional 20-week single group follow-up
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breathing retraining and advice on physical activity (Experimental): 5 minutes of daily diaphragma breathing training, three times per day for 4 weeks
  Interventions: Other: Breathing training; Other: Standrad advice about physical activity
- Standard advice about physical activity (Active Comparator): Written and oral advice about physical activity at baseline
  Interventions: Other: Standrad advice about physical activity

INTERVENTIONS:
Other: Breathing training — Home-based breathing training with written and oral instructions performed 3 x 5 minutes per day for 4 weeks.
  Arms: Breathing retraining and advice on physical activity
Other: Standrad advice about physical activity — Written, standard advice about physical activity at baseline

SUMMARY:
Many children and adolescents with asthma have dysfunctional breathing, e.g. they use mainly upper chest muscles to breath and do not engage the diaphragma muscle when breathing. This can lead to a variety of breathin problems such as dizzyness, muscle tension, and limitations in ability to be physically active. As of today there is no guidelines for treatment or follow-up for these patients and there are very few well-perfomed studies evaluating if breathin retraining can improve breathing pattern.

The aim of this study is to examine the effects of breathing training and advice on physical activity compared to only advice on physical activity in children and adolescents with asthma. The primary outcome is quality of life and secondary outcomes are dysfunctional breathing, asthma control, physical activity level and spirometry changes.

This randomized controlled trial.

Patients are identified at the paediatric lung clinic at Karolinska University Hospital, and patients aged 10-17 years who are reffered to see a physiotherapist for spirometry and exercise testing who have with asthma who have dysfunctional breathing are invited to participate.

Assessments include the Paediatric Asthma Quality of Life Questionnaire, Parent Asthma Quality of Life Questionnaire, The Paediatric Nijmegen Questionnaire assessing symtpoms associated to dysfunctional breathing, the Childhood Asthma control test or the adult asthma control test. These questionnaires as completed by patients with or without their parents depending on their age at baseline, and after 4 weeks, 12 weeks and 24 weeks. At baseline and after 4 weeks an exercise tolerance test of 8 minutes performed on a treadmill and spirometry are performed.

Interventions:

Acitve intervention means diaphragmal breathing training 5 days a week for

DETAILED DESCRIPTION:
Study Protocol for ClinicalTrials.gov

Study Title Effects of Breathing Technique Training and Physical Activity Counseling on Quality of Life, Symptoms, Asthma Control, and Physical Activity in Children and Adolescents With Asthma: A Randomized Controlled Trial

Brief Summary This randomized controlled trial aims to evaluate the effects of training in low-costal and diaphragmatic breathing techniques combined with counseling on physical activity according to FYSS, compared with standard care-physical activity counseling according to FYSS alone-on quality of life, symptoms related to dysfunctional breathing, asthma control, and physical activity levels in children and adolescents with asthma.

Approximately 70 patients referred to a physical therapist at Karolinska University Hospital (Huddinge and Solna) will be invited to participate over one year. Participants will be randomized to either (1) an intervention group receiving extended physiotherapy including breathing training, inhalation technique, and individualized physical activity advice, or (2) a control group receiving standard physical activity recommendations according to FYSS.

The primary outcome is health-related quality of life measured by the Pediatric Asthma Quality of Life Questionnaire (PAQLQ).

Detailed Description This study investigates whether adding structured breathing training to standard physical activity recommendations improves quality of life, dysfunctional breathing symptoms, asthma control, and physical activity levels among children and adolescents aged 10-17 with atopic and/or exercise-induced asthma.

Participants randomized to the intervention group will receive training in low-costal/diaphragmatic breathing, individualized physical activity advice, and inhalation technique training. Diaphragmatic breathing will be practiced 3 times per day for 3-5 minutes. The control group will receive standard physical activity advice based on FYSS guidelines.

Measurements will be taken before and after a 4-week intervention, and at 12- and 24-week follow-ups. Independent physiotherapists at each site will perform all assessments.

Study Design Study Type: Interventional (Clinical Trial) Allocation: Randomized Intervention Model: Parallel Assignment Masking: Single-blinded (Outcome Assessors) Primary Purpose: Treatment Estimated Enrollment: 63 participants Study Duration: 24 weeks follow-up Study Sites: Karolinska University Hospital, Huddinge and Solna

Interventions Intervention Group: Breathing Training + Physical Activity Counseling

* Low-costal/diaphragmatic breathing training (3×/day, 3-5 min)
* Inhalation technique training
* Individualized physical activity advice according to FYSS

Control Group: Standard Physical Activity Counseling (FYSS)

* Aerobic and muscle-strengthening recommendations
* For exercise-induced symptoms: ICS, bronchodilators, gradual warm-up

Outcome Measures Primary Outcome: PAQLQ Secondary Outcomes: Nijmegen Questionnaire, Actigraph accelerometry, ACT, spirometry, treadmill test.

Eligibility Criteria Inclusion: Age 10-17, diagnosis of atopic and/or exercise-induced asthma, referred to physiotherapy.

Exclusion: Completely symptom-free patients.

Study Procedures Baseline: PAQLQ, ACT, Nijmegen Questionnaire, Spirometry, Exercise Test, Accelerometer (14 days).

Intervention Period: 4 weeks. Follow-ups: Week 4, 12, 24.

ELIGIBILITY:
Inclusion Criteria:

* Age 10-17, diagnosis of atopic and/or exercise-induced asthma, referred to physiotherapy.

Exclusion Criteria:

* Completely symptom-free patients, not understanding Swedish language

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2024-08-30 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Paediatric Asthma Quality of Life Questionnaire | Change from baseline in quality of life at 4 weeks. Follow-up at 12 and 24 weeks
  Self-reported quality of life in three domains; Asthma symptoms, Activity limitation and Emotional. Contains 32 items. Completed on paper.
Paediatric Asthma Quality of Life Questionnaire | Assessed at baseline, after 4 weeks of intervention, at 12 weeks and 24 weeks follow-up
  Self-reported quality of life in three domains - symptoms, activity limitation and emotional

SECONDARY OUTCOMES:
Paediatric Nijmegen Questionnaire | Change from baseline in breathing problems at 4 weeks, with follow-up at 12 and 24 weeks
  A newly validated questionnaire to assess symptoms related to dysfunctional breathing for children and adolescents with or with out asthma. Includes 16 items. Based on the original adult Nijmegen Questionnaire.
Saltin-Grimby Physical Activity Scale | Changes from baseline in physical activity levels at 4 weeks with follow-up at 12 and 24 weeks
  Self-reported physical activity level.
Childhood / Adult Asthma Control Test (c-ACT / ACT) | Changes from baseline after 4 weeks of intervention, follow-up at 12 and 24 weeks
  Self-reported control of different asthma signs, 10 imems

CONTACTS AND LOCATIONS:
Overall Officials: Helene Alexanderson, Associate professor, PhD, RPT, Principal Investigator — Medical Unit Allied Health Professionals, Karolinska University Hospital, Stockholm, sweden
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
This is not a a clinical trial investigating safety or effects of a drug and is not funded or organized by NIH. However, we want to share our dataset and statistical analysis accoring to guidelines by the scientific journal who accepts our manuscripts. We would also consider to share results on clincialtrials.gov.

REFERENCES:
- [Background] Juniper EF, Guyatt GH, Cox FM, Ferrie PJ, King DR. Development and validation of the Mini Asthma Quality of Life Questionnaire. Eur Respir J. 1999 Jul;14(1):32-8. doi: 10.1034/j.1399-3003.1999.14a08.x. PMID 10489826
- [Background] Juniper EF, Guyatt GH, Feeny DH, Griffith LE, Ferrie PJ. Minimum skills required by children to complete health-related quality of life instruments for asthma: comparison of measurement properties. Eur Respir J. 1997 Oct;10(10):2285-94. doi: 10.1183/09031936.97.10102285. PMID 9387955
- [Background] van Dixhoorn J, Duivenvoorden HJ. Efficacy of Nijmegen Questionnaire in recognition of the hyperventilation syndrome. J Psychosom Res. 1985;29(2):199-206. doi: 10.1016/0022-3999(85)90042-x. PMID 4009520
- [Background] Thomas M, McKinley RK, Freeman E, Foy C, Prodger P, Price D. Breathing retraining for dysfunctional breathing in asthma: a randomised controlled trial. Thorax. 2003 Feb;58(2):110-5. doi: 10.1136/thorax.58.2.110. PMID 12554890
- [Background] Agache I, Ciobanu C, Paul G, Rogozea L. Dysfunctional breathing phenotype in adults with asthma - incidence and risk factors. Clin Transl Allergy. 2012 Sep 19;2(1):18. doi: 10.1186/2045-7022-2-18. PMID 22992302
- [Background] Hepworth C, Sinha I, Saint GL, Hawcutt DB. Assessing the impact of breathing retraining on asthma symptoms and dysfunctional breathing in children. Pediatr Pulmonol. 2019 Jun;54(6):706-712. doi: 10.1002/ppul.24300. Epub 2019 Apr 1. PMID 30938089
- [Background] Merikallio VJ, Mustalahti K, Remes ST, Valovirta EJ, Kaila M. Comparison of quality of life between asthmatic and healthy school children. Pediatr Allergy Immunol. 2005 Jun;16(4):332-40. doi: 10.1111/j.1399-3038.2005.00286.x. PMID 15943597
- [Background] Bateman ED, Hurd SS, Barnes PJ, Bousquet J, Drazen JM, FitzGerald JM, Gibson P, Ohta K, O'Byrne P, Pedersen SE, Pizzichini E, Sullivan SD, Wenzel SE, Zar HJ. Global strategy for asthma management and prevention: GINA executive summary. Eur Respir J. 2008 Jan;31(1):143-78. doi: 10.1183/09031936.00138707. PMID 18166595